CLINICAL TRIAL: NCT04399187
Title: Clinical Effects of Adjunctive Local Sodium Hypochlorite Gel in Minimally Invasive Non Surgical Debridement (MINSD) of Periodontal Pockets. A 6-month Randomized Controlled Clinical Trial
Brief Title: Adjunctive Local Sodium Hypochlorite Gel in Non Surgical Periodontal Debridement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Messina (Other)
Responsible Party: Principal Investigator, Gaetano Isola, DDS, PhD, Researcher, University of Messina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 16-18
Record Dates: First submitted 2020-05-13; First posted 2020-05-22 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- scaling and root planing, Sodium hypochlorite gel application (Experimental): Periodontal pockets > 5 mm in patients of test group were treated by scaling and root planing and Sodium hypochlorite gel application
  Interventions: Drug: Sodium hypochlorite gel application
- scaling and root planing alone (Placebo Comparator): scaling and root planing alone was performed
  Interventions: Drug: Sodium hypochlorite gel application

INTERVENTIONS:
Drug: Sodium hypochlorite gel application — Patients treated by scaling and root planing and Sodium hypochlorite gel application, meanwhile in patients of control group scaling and root planing alone was performed.
  Other Names: Gel application

SUMMARY:
The aim of this study was to assess the efficacy of minimally invasive nonsurgical debridement (MINSD) of periodontal pockets with or without local amino acid buffered sodium hypochlorite (NaOCl) gel application after 6 months follow-up.

DETAILED DESCRIPTION:
Forty periodontal compromised patients were randomly allocated in two groups. Periodontal pockets > 5 mm in patients of test group were treated by MINSD and NaOCl gel application, meanwhile in patients of control group MINSD alone was performed. Full-mouth plaque score (FMPS) , Full-mouth bleeding score (FMBS), probing depth (PD), clinical attachment level (CAL) and gingival recession (GR) were assessed at baseline and after 6 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with periodontitis;
* Age > 18 years old;
* Patients with at least 10 teeth for arch;
* Presence at least of two teeth with PD > 5 mm for quadrant;
* Single-rooted and multi-rooted teeth;

Exclusion Criteria:

* Patients with systemic diseases;
* Pregnant or lactating;
* Tobacco smokers (> 10 cigarettes/day);
* Previous periodontal treatment in the last 2 years;
* Prolonged antibiotic treatment or anti-inflammatory treatment within 6 months prior to periodontal therapy;
* Furcation involvement;
* Acute periodontal or endodontic abscess;
* Third molars

Ages: 32 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
Probing depth changes | 6-months
  Changes over time in probing depth millimiters

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Isola, Study Chair — University of Messina
Locations (1):
- University of Messina, Messina, Italy

IPD SHARING:
Plan to Share IPD: Yes
Sharing study results
Supporting Information: Study Protocol
Time Frame: 6-months
Access Criteria: University website and pubmed